CLINICAL TRIAL: NCT06656000
Title: Digital Analysis of Mesiodistal Crown Width of Permanent Teeth in a Group of Egyptian Children : a Cross Sectional Pilot Study
Brief Title: Digital Analysis of Mesiodistal Tooth Width
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Toqa Hisham Fathy, Principal investigator, Cairo University
Other Study IDs: digital analysis of M--D width
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Measurement of Crown Width of Permanent Teeth
Keywords: Tooth size, mesiodistal width, Egyptian children.

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week

SUMMARY:
the goal of this cross-sectional study is to determine the digital permanent crown tooth width

DETAILED DESCRIPTION:
using digital intra oral scanning to measure the permanent tooth mesiodistal dimension

ELIGIBILITY:
Inclusion Criteria:

* Children range age 12-15 years old.
* Complete set of permanent dentitions with intact marginal ridges.
* Fully erupted teeth to the occlusal plane.
* Normal occlusion without crowding, rotation, Spacing.
* Healthy children with no systemic diseases.

Exclusion Criteria:

* Buildups, Crowns, onlays, class II restorations that affect a tooth mesiodistal
* diameter.
* Congenital defects or deformed teeth or congenital missing Teeth.
* Obvious interproximal or occlusal wear of teeth.
* Anterior teeth fractures.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Healthy Children 12-15 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Digital mesioidistal crown width of permanent anterior and Posterior teeth | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry , Cairo University, Cairo, Egypt